CLINICAL TRIAL: NCT02975050
Title: Vital Signs Validation Study of the μ-Cor System (ViVUS Validation)
Acronym: ViVUS
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-KM-001
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Health Volunteer Validation Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Side location: u-Cor device will be applied on side location
  Interventions: Other: Location
- Front location: u-Cor device will be applied on front location
  Interventions: Other: Location

INTERVENTIONS:
Other: Location

SUMMARY:
This study has the following objective:

• To validate the capability of the μ-Cor System to monitor ECG, Heart Rate (HR), Respiration Rate (RR), Posture and Activity in healthy human subjects.

The μ-Cor validation will be demonstrated at two body locations:

1. Side location (below left armpit) for study arm 1, and
2. Front location (upper left chest) for study arm 2 An FDA-cleared comparator device will be used to support the validation of the study device.

DETAILED DESCRIPTION:
This study has the following objective:

• To validate the capability of the μ-Cor System to monitor ECG, Heart Rate (HR), Respiration Rate (RR), Posture and Activity in healthy human subjects.

The μ-Cor validation will be demonstrated at two body locations:

1. Side location (below left armpit) for study arm 1, and
2. Front location (upper left chest) for study arm 2 An FDA-cleared comparator device will be used to support the validation of the study device.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 21 years of age or older.
* Subject is willing and able to sign the Informed Consent Form.
* Subject is healthy, able and willing to complete all the preparation steps and study procedures.

Exclusion Criteria

* Female subject with a known pregnancy or unsure about pregnancy status.
* Subjects with allergies and/or skin sensitivities to electrode hydrogel and/or acrylic based adhesive.
* Subjects with skin breakdown in areas where device placement is required.
* Subjects with chronic lung disease or asthma.
* Subjects with a history of cardiovascular diseases.
* Subjects who are diabetic.
* Subjects living with kidney failure or dialysis.
* Subjects with a history of liver failure.
* Subjects with any known malignancy (i.e. cancer patients).
* Subjects with implanted devices in the thoracic region

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Respiratory rate | Immediately
  The difference between the μCor RR and the comparator RR will be lower than 2.8bpm (STD).
Posture | Immediately
  90% agreement between the positions (supine / reclined / upright) derived from μCor reporting and the known position
Activity | Immediately
  μCor output is provided as "active" and "not active". 90% correct classification of activity will be required of recordings.
Heart Rate | Immediately
ECG | Immediately

IPD SHARING:
Plan to Share IPD: No